CLINICAL TRIAL: NCT00421928
Title: A Randomized Double-Blind, Placebo- and Active-Control, Parallel-arm, Phase III Trial With Controlled Adjustment of Dose to Evaluate the Efficacy and Safety of CG5503 Extended-Release (ER) in Patients With Moderate to Severe Chronic Pain Due to Osteoarthritis of the Knee
Brief Title: Tapentadol (CG5503)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Grünenthal GmbH (Industry)
Responsible Party: Director, Clinical Leader, Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR013402; R331333PAI3008 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.); KF11 (Other: Grunenthal GMBH)
Record Dates: First submitted 2007-01-12; First posted 2007-01-15 (Estimated); Results first posted 2010-04-23 (Estimated); Last update posted 2012-04-18 (Estimated); Status verified 2012-04

CONDITIONS: Osteoarthritis, Knee; Pain
Keywords: Chronic Pain; Osteoarthritis, Knee; tapentadol; Pain Assessment
MeSH Terms: conditions — Osteoarthritis, Knee; Pain; Chronic Pain | interventions — Oxycodone; Tapentadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 001 (Experimental): tapentadol (CG5503) 50 100 150 200 250mg twice a day (BID) during 15 weeks
  Interventions: Drug: tapentadol (CG5503)
- 002 (Active Comparator): oxycodone 10 20 30 40 50mg twice a day (BID) during 15 weeks
  Interventions: Drug: oxycodone
- 003 (Placebo Comparator): placebo matching placebo twice a day (BID) during 15 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: oxycodone — 10, 20, 30, 40, 50mg twice a day (BID) during 15 weeks
  Arms: 002
Drug: placebo — matching placebo twice a day (BID) during 15 weeks
  Arms: 003
Drug: tapentadol (CG5503) — 50, 100, 150, 200, 250mg twice a day (BID) during 15 weeks
  Arms: 001

SUMMARY:
The purpose of this trial is to evaluate the effectiveness (level of pain control) and safety of orally administered tapentadol (CG5503) Extended Release (ER) (base) at doses of 100-250 mg twice daily in patients with moderate to severe chronic pain due to osteoarthritis of the knee, in comparison with placebo and Oxycodone Controlled Release (CR).

DETAILED DESCRIPTION:
The primary objective of this randomized (study medication assigned to patients by chance), double-blind (neither patient nor investigator knows the study medication) , phase III, placebo and active controlled trial is to evaluate the efficacy and safety of orally administered tapentadol (CG5503) Extended Release (ER) (base) at doses of 100-250 mg twice daily in patients with moderate to severe chronic pain from osteoarthritis (OA) of the knee. The study is being conducted for registration and approval of tapentadol (CG5503) in the US and outside the US. The trial will consist of five periods: screening (to assess eligibility) , washout (3-7 days with determination of a baseline pain intensity), titration (of dose over 3 weeks to the optimal individual level) , maintenance (investigational drug intake for 12 weeks with adjustments allowed), and follow-up (2 weeks post treatment discontinuation). The study hypothesis is that the study drug will be more effective than placebo in reducing patients pain intensity. The Secondary objectives include the collection of pharmacokinetic (related to how the body uses the drug) information for dose verification. The trial objectives will be assessed by comparing the baseline pain level to the level of week 12 of the maintenance phase. This will be done by looking at the patient's pain diary information. Titrate tapentadol (CG5503) ER (extended release) 50mg to patient's optimal dose ranging between 100mg and 250mg twice a day; Oxycodone CR (controlled release) 10mg to 50mg twice a day; Placebo (no active ingredients). All doses of trial treatment will be taken orally with approximately 120 mL of water with or without food for a maximum timeframe of 15 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with osteoarthritis of the knee based on the American College of Rheumatology (ACR) criteria and functional capacity class of I-III
* patients taking analgesic medications for at least 3 months prior to screening and/or dissatisfied with their current therapy
* Patients requiring opioid treatment must be taking daily doses of opioid-based analgesic, equivalent to <160 mg of oral morphine
* baseline score of greater than or equal to 5 on an 11-point numerical rating scale, calculated as the average pain intensity during the last 3 days prior to randomization.

Exclusion Criteria:

* History of alcohol and/or drug abuse in Investigator's judgement
* history of significant liver insufficiency
* chronic hepatitis B or C, or HIV, presence of active hepatitis B or C within the past 3 months
* life-long history of seizure disorder or epilepsy
* history of malignancy within past 2 years, with exception of basal cell carcinoma that has been successfully treated
* uncontrolled hypertension
* patients with severely impaired renal function
* patients with moderate to severly impaired hepatic function or with laboratory values reflecting inadequate hepatic function

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1030 (Actual)
Dates: Start 2007-01; Primary Completion 2008-07 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Etropolski M, Kuperwasser B, Flugel M, Haufel T, Lange B, Rauschkolb C, Laschewski F. Safety and tolerability of tapentadol extended release in moderate to severe chronic osteoarthritis or low back pain management: pooled analysis of randomized controlled trials. Adv Ther. 2014 Jun;31(6):604-20. doi: 10.1007/s12325-014-0128-6. Epub 2014 Jul 2. PMID 24985410
- [Derived] Biondi DM, Xiang J, Etropolski M, Moskovitz B. Evaluation of blood pressure and heart rate in patients with hypertension who received tapentadol extended release for chronic pain: a post hoc, pooled data analysis. Clin Drug Investig. 2014 Aug;34(8):565-76. doi: 10.1007/s40261-014-0209-y. PMID 24916058
- [Derived] Etropolski M, Lange B, Goldberg J, Steup A, Rauschkolb C. A pooled analysis of patient-specific factors and efficacy and tolerability of tapentadol extended release treatment for moderate to severe chronic pain. J Opioid Manag. 2013 Sep-Oct;9(5):343-56. doi: 10.5055/jom.2013.0177. PMID 24353047
- [Derived] Merchant S, Provenzano D, Mody S, Ho KF, Etropolski M. Composite measure to assess efficacy/gastrointestinal tolerability of tapentadol ER versus oxycodone CR for chronic pain: pooled analysis of randomized studies. J Opioid Manag. 2013 Jan-Feb;9(1):51-61. doi: 10.5055/jom.2013.0147. PMID 23709304
- [Derived] Afilalo M, Morlion B. Efficacy of tapentadol ER for managing moderate to severe chronic pain. Pain Physician. 2013 Jan;16(1):27-40. PMID 23340531
- See also: A Randomized Double-Blind, Placebo & Active-Control, Parallel-Arm Phase 3 Study With Controlled Dose Adjustment to Evaluate the Efficacy and Safety of Tapentadol Extended-Release (ER) in Subjects With Moderate to Severe Chronic Pain Due to OA of the Knee — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=69&filename=CR013402_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period for this out-patient, multicenter study occurred between 07 February 2007 and 15 July 08.
Pre-assignment Details: The study consisted of a screening period (duration up to 14 days), a washout period (duration 3 to 7 days), a double-blind active treatment period with titration period (duration 3 weeks) and maintenance period (duration 12 weeks)
Groups:
- Tapentadol (CG5503): Tapentadol(CG5503) extended release (ER) 100-250mg twice daily (BID)
- Oxycodone: oxycodone controlled release (CR)20-50mg twice daily (BID)
- Placebo: Matching Placebo twice daily (BID)
Period: Overall Study
Arm/Group | Tapentadol (CG5503) | Oxycodone | Placebo
Started | 344 (2 randomly assigned to this treatment group did not receive drug) | 342 (2 randomly assigned to this treatment group did not receive drug. One subject was enrolled twice.) | 337 (2 randomly assigned to this treatment group did not receive drug)
Completed | 181 | 118 | 203
Not Completed | 163 | 224 | 134
Not completed — Adverse Event | 61 | 140 | 22
Not completed — Lost to Follow-up | 5 | 0 | 3
Not completed — Withdrawal by Subject | 50 | 48 | 43
Not completed — Lack of Efficacy | 15 | 7 | 35
Not completed — Study drug non-compliant | 6 | 7 | 4
Not completed — All other | 26 | 21 | 27
Not completed — Death | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tapentadol (CG5503) | Oxycodone | Placebo | Total
Number analyzed (Participants) | 344 | 342 | 337 | 1023
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 249 | 249 | 260 | 758
  >=65 years | 95 | 93 | 77 | 265
Age Continuous [Mean (Standard Deviation); unit: years] | 58.4 (10.09) | 58.2 (10.29) | 58.2 (9.15) | 58.3 (9.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 216 | 202 | 200 | 618
  Male | 128 | 140 | 137 | 405

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of the Average Pain Intensity Based on an 11-point Numerical Rating Scale(NRS) Over the Last Week of the Maintenance Period at Week 12.
Description: For this twice daily pain assessment, the subjects were to indicate the level of pain experienced over the previous 12 hours on an 11-point Numerical Rating Scale (NRS) where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine".
Time Frame: Baseline and 12 weeks (Primary endpoint is the average pain intensity score during the last week of the maintenance period).
Population: Intent-to-treat (ITT) population. Last observation carried forward (LOCF) was used to impute pain score after discontinuation
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tapentadol (CG5503) | Oxycodone | Placebo
Number analyzed (Participants) | 344 | 342 | 337
Scores on a scale | -3.0 (2.39) | -2.6 (2.38) | -2.2 (2.54)
Statistical Analysis 1: Comparison: Tapentadol (CG5503) vs Placebo; The primary null hypothesis to be tested for the study was that the tapentadol ER group was not different from the placebo group for the primary endpoint. Assuming the mean treatment group difference of 0.7 with an SD of 2.7, 314 subjects per treatment group were estimated to provide 90% power to show that the tapentadol ER group was statistically different from placebo at an alpha level of 0.05. The total number of subjects to be randomly assigned to a treatment group for the study was 942; Test type: Superiority or Other; p < 0.05, ANCOVA; Analysis of covariance (ANCOVA) model was used with treatment and pooled analysis center as factors and baseline pain intensity score as a covariate; Mean Difference (Final Values) = -0.7, 95% CI [-1.04 to -0.33], Standard Error of Mean 0.18

2. Secondary Outcome: Change From Baseline in Western Ontario McMaster Questionnaire (WOMAC) Assessing Pain, Disability and Joint Stiffness of the Knee Over the Last Week of the Maintenance Period at Week 12
Description: Change from baseline to Week 12 of WOMAC Global Score: WOMAC is measure with a Likert ordinal scale from 0-4 with lower scores indicating lower levels of symptoms or physical disability
Time Frame: Baseline and 12 week endpoint
Population: Intent To Treat (ITT), observed cases analysis conducted, no imputation performed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tapentadol (CG5503) | Oxycodone | Placebo
Number analyzed (Participants) | 149 | 92 | 158
Scores on a scale | -1.2 (0.82) | -1.1 (0.87) | -0.9 (0.84)

3. Secondary Outcome: Change From Baseline in Sleep Latency Time in Hours Over the Last Week of the Maintenance Period at Week 12.
Description: A Sleep Questionniare addressed the following question: "How long after bedtime/lights out did you fall asleep last night (hours)?" 12 week endpoint-mean changes from baseline at endpoint for sleep latency. Decrease in time(hours) indicates improvement.
Time Frame: Baseline and 12 week endpoint
Population: ITT
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Tapentadol (CG5503) | Oxycodone | Placebo
Number analyzed (Participants) | 339 | 337 | 331
Hours | 0.2 (2.8) | 0.1 (1.81) | 0.3 (2.72)

4. Secondary Outcome: Percentage of Patients Who Reported Very Much Improved or Much Improved From Baseline in Patient Global Impression of Change Over the Last Week of the Maintenance Period at Week 12
Description: Ordinal measure indicating change from start of treatment (on a scale of 7 = Very much worse to 1 = Very much improved)
Time Frame: Baseline and 12 week endpoint
Population: ITT
Measure: Number; unit: percentage of participants
Arm/Group | Tapentadol (CG5503) | Oxycodone | Placebo
Number analyzed (Participants) | 317 | 308 | 309
percentage of participants | 51.1 | 37.7 | 32.4

5. Secondary Outcome: Distribution of Time to Treatment Discontinuation Due to Lack of Efficacy
Description: The median time to treatment discontinuation due to lack of efficacy from baseline to endpoint
Time Frame: Baseline to 12 weeks
Population: ITT: The results for median and interquartile ranges were not estimable because insufficient number of subjects discontinued due to lack of efficacy to estimate the values.
Measure: Number; unit: median time
Arm/Group | Tapentadol (CG5503) | Oxycodone | Placebo
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Change From Baseline in EuroQol-5 (EQ-5D) Health Status Index to Week 12
Description: Change from baseline to end point in EuroQol-5 (EQ-5D) Dimension Questionnaire. A higher score indicates an improvement in health in the Health Status Index. The EQ-5D is a five dimensional health state classification. Each dimension is assessed on a 3-point ordinal scale (1=no problems, 2=some problems, 3=extreme problems). The responses to the five EQ-5D dimensions were scored using a utility-weighted algorithm to derive an EQ-5D health status index score between 0 to 1, with 1.00 indicating "full health" and 0 representing dead
Time Frame: Baseline and 12 week endpoint
Population: ITT
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Tapentadol (CG5503) | Oxycodone | Placebo
Number analyzed (Participants) | 344 | 342 | 337
scores on a scale | 0.6 (0.26) | 0.5 (0.28) | 0.5 (0.29)

7. Secondary Outcome: Change From Baseline in Responder Analysis 50% Improvement to Week 12
Description: Defined by the percentage of subjects achieving at least 50% improvement from baseline in the primary endpoint based on the 11-point NRS at week 12. For this twice daily pain assessment, the subjects were to indicate the level of pain experienced over the previous 12 hours on an 11-point Numerical Rating Scale (NRS) where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine".
Time Frame: Baseline and Week 12
Population: ITT. Subjects who discontinued from the study were considered non-responders.
Measure: Number; unit: Percentage of participants
Arm/Group | Tapentadol (CG5503) | Oxycodone | Placebo
Number analyzed (Participants) | 344 | 342 | 337
Percentage of participants | 32.0 | 17.3 | 24.3

ADVERSE EVENTS:
Time Frame: All adverse events were reported from the time a signed and dated informed consent was obtained throughout the follow-up phase of the study. Serious adverse events were collected for 30 days after the last dose of study drug.
Arm/Group | Tapentadol (CG5503) | Oxycodone | Placebo
Serious Adverse Events (participants affected / at risk) | 4/344 | 10/342 | 6/337
Other Adverse Events (participants affected / at risk) | 200/344 | 269/342 | 134/337
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tapentadol (CG5503) (N=344) | Oxycodone (N=342) | Placebo (N=337)
Myocardial Infarction (Cardiac disorders) | 0 | 1 | 1
Cardiac Failure Congestive (Cardiac disorders) | 1 | 0 | 0
Angina Pectoris (Cardiac disorders) | 0 | 1 | 0
Atrial Flutter (Cardiac disorders) | 0 | 1 | 0
Meniere's Disease (Ear and labyrinth disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Pyelonephritis Acute (Infections and infestations) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal Mass (Gastrointestinal disorders) | 0 | 1 | 0
Drug Withdrawal Syndrome (General disorders) | 0 | 1 | 0
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Embolic Stroke (Nervous system disorders) | 0 | 0 | 1
Confusional State (Psychiatric disorders) | 0 | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 0 | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Spinal Fusion Surgery (Surgical and medical procedures) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tapentadol (CG5503) (N=344) | Oxycodone (N=342) | Placebo (N=337)
Nausea (Gastrointestinal disorders) | 74 | 125 | 23
Constipation (Gastrointestinal disorders) | 65 | 126 | 22
Dry Mouth (Gastrointestinal disorders) | 22 | 15 | 8
Vomiting (Gastrointestinal disorders) | 18 | 61 | 11
Diarrhoea (Gastrointestinal disorders) | 16 | 17 | 20
Dizziness (Nervous system disorders) | 61 | 65 | 16
Headache (Nervous system disorders) | 51 | 50 | 56
Somnolence (Nervous system disorders) | 37 | 67 | 14
Fatigue (General disorders) | 37 | 35 | 15
Pruritus (Skin and subcutaneous tissue disorders) | 24 | 43 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 6 | 17
Back Pain (Musculoskeletal and connective tissue disorders) | 7 | 5 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less